CLINICAL TRIAL: NCT03602547
Title: Phase II Clinical Study of CM082 Combined With JS001 in the Treatment of Advanced Mucosal Melanoma.
Brief Title: Study of the Combination of CM082 With JS001 in Patients With Advanced Mucosal Melanoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-II-202
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Mucosal Melanoma
MeSH Terms: interventions — vorolanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM082 plus JS001 (Experimental): Patients who meet the enrollment criteria will receive CM082 tablets 200mg once daily (qd) orally (taken within half an hour after daily breakfast) in combination with JS001 (3mg/kg, once every 2 weeks, q2w), every 28 days A treatment cycle until the disease progresses, the toxicity is intolerable, the investigator or subject decides to withdraw, loses to follow up, starts using other anti-tumor treatments or dies.
  Interventions: Drug: CM082 plus JS001

INTERVENTIONS:
Drug: CM082 plus JS001 — CM082：200mg once a day (qd) orally (taken within half an hour after breakfast). JS001 :An intravenous infusion of a solution having a concentration of 1-10 mg/ml was prepared with 0.9% physiological saline, and administered once every two weeks. Using an inline filter (0.2 or 0.22 μm), the drug was diluted with physiological saline and intravenously administered within 60 minutes.

SUMMARY:
This study was a one-arm, single-center, phase II clinical study. Patients who meet the enrollment criteria will receive CM082 tablets 200mg once daily (qd) orally (taken within half an hour after daily breakfast) in combination with JS001 (3mg/kg, once every 2 weeks, q2w), every 28 days a treatment cycle until the disease progresses , the toxicity is intolerable, the investigator or subject decides to withdraw, loses to follow up, starts using other anti-tumor treatments or dies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of recurrence after surgery, inoperable resection or metastasis advanced mucinous melanoma (III/IV period).
* Has not received any systemic anti-tumor medication (previously adjuvant or neoadjuvant therapy is required, but the treatment should be completed for at least 4 weeks prior to the first dose of study drug, and all related toxicity events have returned to normal or no more than Grade I of CTCAE 4.03, except for hair loss).
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1.
* Life expectancy of at least 12 weeks.
* All patients should provid tumor tissue specimens (preferably fresh tissue specimens) for PD-L1 expression analysis prior to enrollment.
* There is at least one measurable lesion according to the RECIST 1.1 standard and the lesion has not received radiotherapy.
* Patients may have a history of brain/mesis metastases, but must undergo topical treatment(surgery/radiotherapy) and be clinically stable for at least 3 months prior to the start of the study .If orticosteroids have been used before, they should be discontinued for at least 2 weeks before the first dose of study drug.
* The level of organ function must meet the following requirements (7 days before the first dose of study drug):

  * Bone marrow: Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L, platelet (PLT) ≥ 100 × 109 / L, hemoglobin (HB) ≥ 9g / dL (no blood transfusion or receiving blood components within 14 days before detection);
  * Liver: serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal（ULN）, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5*ULN (if liver metastasis, AST, ALT allowed) ≤ 5 *ULN);
  * Serum creatinine ≤ 1.5*ULN and endogenous creatinine clearance ≥ 50mL / min (Cockcroft-Gault formula);
  * Well-controlled hypertensive patients can be enrolled;
  * International normalized ratio (INR), activated partial thromboplastin time (aPTT) ≤ 1.5 *ULN for patients who have not received anticoagulant therapy; patients who receive anticoagulant therapy should be treated within the requirements of label
  * Urine protein ≤ 1+, if urine protein > 1+, 24 hours urine protein measurement is required, the total amount of which needs ≤ 1 gram;
  * FT3, FT4, TSH normal or abnormal has no clinical significance;
  * The heart function is normal, that is, the electrocardiogram is normal or abnormal has no clinical significance. The echocardiography shows that the left ventricular ejection fraction (LVEF) is greater than 50%.
* Serum pregnancy test results must be negative within 7 days prior to the first dose of the test drug for women of childbearing age; males with fertility or women who are at risk of pregnancy must use highly effective methods of contraception throughout the trial (eg oral contraceptives, pIntrauterine device, controlled libido or barrier contraceptive method combined with spermicide), and continued contraception for 12 months after the end of treatment.
* Ability to understand the nature of this trial and give written informed consent.Willingness and ability to comply with trial and follow-up procedures

Exclusion Criteria:

* Patients who have previously received anti-PD-1, anti-PD-L1, anti-PD-L2 therapy, or VEGFR TKI therapy.
* Patients currently receiving anti-tumor treatment
* Patients who participated in or were participating in other drug/therapy clinical trials within 4 weeks prior to the first dose of the study drug.
* Patients who received large surgery within 4 weeks before the first dose of the test drug or has not recovered from the side effects of this operation, received live vaccination or immunotherapy within 4 weeks before the first dose of the test drug, and radiotherapy was performed within 2 weeks.

In the past 5 years, there have been history of malignant tumors other than mucosal melanoma, except for cured skin basal cell carcinoma, cutaneous squamous cell carcinoma, early prostate cancer, and cervical carcinoma in situ.

* Hematopoietic stimulating factors were received within 1 week prior to the first dose of the study drug, such as granulocyte colony-stimulating factor (G-CSF) and erythropoietin.
* HIV antibody or Treponema pallidum antibody test results are positive.
* If HBsAg or HBcAb is positive, HBV DNA should be tested.Patients should be excluded if the measurement is above the upper limit of the normal range.If HCV antibody is positive, HCV DNA should be tested.Patients should be excluded if the measurement is above the upper limit of the normal range.
* Those known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components; those known to be allergic to CM-082 and any of its excipients.
* A large amount of pleural or ascites with clinical symptoms and requiring symptomatic treatment.
* Active lung disease (eg, interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or a history of active tuberculosis.
* Have any clinical problems out of control, including but not limited to:

  * Persistent or active (severe) infection;
  * Hypertension that is not effectively controlled (blood pressure lasts greater than 150/90mmHg);
  * Diabetes that is not effectively controlled;
  * Heart disease, defined as grade III/IV congestive heart failure or heart block defined by the New York Heart Association
  * Having a history of or suspected of having an autoimmune disease;Having a history of any kind of disease requiring treatment with a steroid/immunosuppressive, such as: pituitary inflammation, colitis, hepatitis, nephritis, hyperthyroidism, Hypothyroidism, etc.;
  * The following situation occurred within 6 months before the first dose:

    * Deep vein thrombosis or pulmonary embolism;
    * myocardial infarction;
    * severe or unstable arrhythmia or angina;
    * percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting;
    * Cerebrovascular accident, transient ischemic attack, and cerebral embolism.
* The patient has any condition that affects the swallowing of the drug, as well as any conditions that affect the course of treatment (absorption, distribution, metabolism, or excretion) of the test drug, including any type of gastrointestinal resection or surgical history.
* Have received a stem cell transplant or an organ transplant.
* Has a history of psychotropic substance abuse which is unable to quit or has a history of mental disorders.
* Patients who need to use during the study or have used or the following drugs within 14 days prior to the first dose: CYP3A4 strong inhibitor or strong inducer; warfarin or any other coumarin derivative anticoagulant.
* The investigator judges other severe, acute or chronic medical illness or laboratory abnormalities that may increase the risk associated with the study or may interfere with the interpretation of the findings.
* The investigator judged that the patient's compliance was poor or that there were other conditions that were not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 12 months
  The proportion of patients with complete remission (CR) and partial remission (PR) in all patients.Disease progression will be evaluated according to Response Evaluation Criteria in Solid Tumors V 1.1.

SECONDARY OUTCOMES:
Disease Control Rate | 12 months
  The proportion of patients with complete remission (CR),partial remission (PR) and stable diseasein(SD) all patients.Disease progression will be evaluated according to Response Evaluation Criteria in Solid Tumors V 1.1 and Immune-related Response Criteria.
Duration of Response | 12 months
  The time interval between the first time of being evaluated as complete response (CR) or partial response (PR) and the first time of being evaluated as progressed disease(PD).Disease progression will be evaluated according to Response Evaluation Criteria in Solid Tumors V 1.1 and Immune-related Response Criteria.
Time to Response | 12 months
  Time from randomization to complete response (CR) or partial response (PR).Disease progression will be evaluated according to Response Evaluation Criteria in Solid Tumors V 1.1 and Immune-related Response Criteria.
Progression-free survival | 12 months
  The internal between the date of randomization and the date of disease progression, unaccepted toxicity, or death
Overall survival | 36 months
  The internal between the date of randomization and the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, M.D, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China